CLINICAL TRIAL: NCT06218238
Title: Do Transfemoral Prostheses With Powered Prosthetic Knee Flexion and Extension Improve Mobility? A Biomechanical Evaluation of the Ossur Power Knee
Brief Title: A Biomechanical Evaluation of the Ossur Power Knee in Persons With Transfemoral Amputation
Acronym: OPKTFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4541-R; RX004541-01A2 (Other Grant/Funding Number: VA RRD)
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Transfemoral Amputation; Limb Loss; Limb Absence
Keywords: amputation; limb loss; limb deficiency; transfemoral; above-knee; prosthesis; knee joint

STUDY DESIGN:
Intervention Model Description: Using a cross-over experimental design, 20 unilateral, transfemoral amputee subjects (10 men and 10 women) will be evaluated in the Jesse Brown VAMC Motion Analysis Research Laboratory (MARL) while wearing the Ossur Power Knee and Ossur Rheo XC. Subjects will be provided a one-month accommodation period wearing each prosthetic knee prior to testing. Prosthetic foot type will be standardized for subjects so they will walk with the same foot while testing each prosthetic knee joint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ossur Power Knee (Experimental): Subjects will be fitted with the Ossur Power Knee, which has powered flexion and extension.
  Interventions: Other: Powered prosthetic knee joint
- Ossur Rheo XC Knee (Active Comparator): Subjects will be fitted with the Ossur Rheo XC Knee, which is a conventional microprocessor-controlled knee joint that modulates the amount of damping during flexion and extension.
  Interventions: Other: Conventional prosthetic knee joint

INTERVENTIONS:
Other: Powered prosthetic knee joint — Subjects will be fitted and trained on the Ossur Power Knee. An accommodation of 1 month will be provided prior to evaluation with the knee joint.
  Arms: Ossur Power Knee
Other: Conventional prosthetic knee joint — Subjects will be fitted and trained on the Ossur Rheo XC Knee. An accommodation of 1 month will be provided prior to evaluation with the knee joint.
  Arms: Ossur Rheo XC Knee

SUMMARY:
Microprocessor-controlled knees (MPKs) do not typically utilize motors to power joint rotation, but they automatically adjust resistance or damping in the joint to improve swing- and/or stance-phase control as appropriate for the prosthesis user during gait. The Ossur Power Knee is the only commercially-available MPK that uses a motor to provide active power generation during walking and other activities. The purpose of this proposed investigation is to perform and compare biomechanical evaluations of the Power Knee and Ossur Rheo XC, a passive MPK, during walking and other activities by prosthesis users. Furthermore, mobility between male and female subjects will be compared to determine if there are differences in prosthetic knee usage on the basis of sex.

DETAILED DESCRIPTION:
The anatomical knee is a complex, polycentric joint characterized by a large range of motion in the sagittal plane and limited mobility in the coronal and transverse planes. The sagittal plane motion is used for progression in stance phase, and limb clearance and advancement in swing. Limb prostheses are intended to restore function and cosmesis in persons with limb loss. The complexity and function of prosthetic components have advanced significantly as technology has improved, but a state-of-the-art artificial limb is still a relatively poor substitute for an anatomical one. Microprocessor-controlled knees (MPKs) do not typically utilize motors to power joint rotation, but they automatically adjust resistance or damping in the joint to improve swing- and/or stance-phase control as appropriate for the user during gait. The Ossur Power Knee, which was first introduced in 2006, is the only MPK that uses a motor to provide active power generation during walking and other activities involving knee flexion and extension. Last year, Ossur released the 3rd generation of its Power Knee and appears to have addressed many of the previous shortcomings in terms of reduced weight, less noise, lower cost and longer battery life. Therefore, the newest version of the Power Knee warrants a fresh evaluation since it is, in essence, substantially different in design and function from previous models.

The purpose of this proposed investigation is to perform biomechanical evaluations of the new Ossur Power Knee during walking and other activities by transfemoral prosthesis users. Using a cross-over experimental design, approximately 20 unilateral, transfemoral amputee subjects (10 men and 10 women) will be evaluated in the Jesse Brown VAMC Motion Analysis Research Laboratory (MARL) while wearing the Ossur Power Knee and Ossur Rheo XC, which is a passive MPK device. Furthermore, the Ossur Power Knee may offer distinct advantages to female prosthesis users, so mobility will be compared between men and women to determine if differences exist on the basis of sex. The specific aims and hypotheses of this project are:

Aim 1: To compare the effects of the Ossur Power Knee and Ossur Rheo XC on the gait of unilateral, transfemoral prosthesis users during level walking. Kinematic and kinetic data will be collected as subjects walk in the MARL. Hypothesis--the active knee flexion and extension provided by the Ossur Power Knee will (1) improve walking performance, and (2) reduce metabolic energy cost during ambulation.

Aim 2: To compare the effects of the Ossur Power Knee and Ossur Rheo XC on stairs, slopes and during sit-to-stand/stand-to-sit activities of unilateral, transfemoral prosthesis users. Kinematic data will be collected as subjects perform these activities. Hypothesis--subjects will have improved performance when using the Ossur Power Knee.

Aim 3: To analyze and compare gender specific data between subjects using the Ossur Power Knee and the Ossur Rheo XC. Hypothesis--male and female subjects will demonstrate substantially different abilities to use the two knee components, indicating that gender specific components should be further investigated and developed. Research focusing on the unique prosthetic needs of women Veterans is currently a special emphasis area of the VA RR&D Service.

Subjects will also be administered questionnaires and provided at-home diaries to document their perceptions of comfort, exertion and stability while using the different prosthetic knee units.

The repeated-measures, cross-over protocol design enables each subject to serve as their own control, and it will be determined whether statistically significant changes occur in their performance measures. A two-way mixed-methods ANOVA will be used to assess the main and interaction effects of sex (male, female) and knee type (Ossur Power Knee, Rheo XC). As a conservative approach, a Bonferroni correction will be used to account for the family-wise Type I error rate because multiple outcomes will be used to address each hypothesis.

Increased understanding about how the Ossur Power Knee affects the abilities of transfemoral prosthesis users will facilitate appropriate component selection by prosthetists and ultimately improve quality of life for prosthesis users.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral, transfemoral amputation (any etiology).
* Age from 45-75 years.
* Residual limb length classified as standard (i.e., medium) to long.
* Prosthesis user for at least 1 year prior to enrolling in the study.
* K3 or K4 level ambulator.
* Good sensation on their residual limb(s) (upon routine clinical examination).
* Good skin integrity upon visual inspection.
* Does not require the use of assistive devices to walk for short distances.
* Not currently taking medications that are known to affect balance or gait.
* Presents with good socket fit based upon a standard assessment by the study prosthetist.

Exclusion Criteria:

* Bilateral amputations
* Individuals with a knee disarticulation

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A total of 10 males and 10 females will be enrolled in this study. Subjects must meet the inclusion/exclusion criteria listed previously.
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Walking speed | To be measured after the 1-month accommodation period of wearing each prosthetic knee component
  Walking speed will be measured as participants walk on level ground at slow, normal and fast speeds.
Metabolic energy cost | To be measured after the 1-month accommodation period of wearing each prosthetic knee component
  The metabolic energy rate will be measured as subjects walk at their freely selected speed on a level treadmill, which will be converted to metabolic energy cost (energy expended per unit distance).
Sit-to-stand/stand-to-sit symmetry | To be measured after the 1-month accommodation period of wearing each prosthetic knee component
  Knee kinematics and load distribution between the sound and prosthetic sides will be measured as participants stand up and sit down in a chair.

SECONDARY OUTCOMES:
Step length | To be measured after the 1-month accommodation period of wearing each prosthetic knee component
  The step lengths of the sound and prosthetic sides will be measured as participants walk on level ground at slow, normal and fast speeds.
Toe clearance during swing phase | To be measured after the 1-month accommodation period of wearing each prosthetic knee component
  Toe clearance during swing phase on the prosthetic side will be measured as participants walk on level ground at slow, normal and fast speeds.
Sound leg loading rate | To be measured after the 1-month accommodation period of wearing each prosthetic knee component
  The sound leg loading rate during walking will be measured as participants walk on level ground at slow, normal and fast speeds.
Kinematics of pelvic motion | To be measured after the 1-month accommodation period of wearing each prosthetic knee component
  Pelvic tilt, rotation and obliquity will be measured as participants walk on level ground at slow, normal and fast speeds.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Gard, PhD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. Results from this study will be freely disseminated via presentations at professional conferences and publications in scientific journals. Additionally, data acquired for this project will be shared with those investigators who make a formal request to the PI and can demonstrate a legitimate and justifiable cause for utilization of such data. All requests for these data will be discussed with the VA scientific program manager.